CLINICAL TRIAL: NCT01213407
Title: First Line Standard Therapy of Glioblastoma Multiforme With or Without add-on Treatment With Trivax, an Anti-tumour Immune Therapy Based on Tumour-lysate Charged Dendritic Cells
Brief Title: Dendritic Cell Cancer Vaccine for High-grade Glioma
Acronym: GBM-Vax
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Activartis Biotech (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: GBM-Vax-TRX2
Record Dates: First submitted 2010-05-28; First posted 2010-10-04 (Estimated); Last update posted 2016-05-19 (Estimated); Status verified 2016-05

CONDITIONS: Glioblastoma Multiforme
Keywords: Dendritic cell; Cancer vaccine; Anti-tumor immune therapy; Interleukine-12; Individualised autologous therapy; Brain cancer; Temozolomide; Radiotherapy; Irradiation; High-grade glioma; Advanced therapy medicinal product ATMP; Somatic cell therapy; Leukocyte apheresis; Neurosurgery; Neurooncology; Neurology; Immunology; Tumor immunology; Transfusion medicine; Monocyte; Killer cell; Cytotoxic T-cell; Cytotoxic T-lymphocyte
MeSH Terms: conditions — Glioblastoma; Brain Neoplasms; Glioma | interventions — Temozolomide; Surgical Procedures, Operative; Radiotherapy

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Standard therapy plus Trivax (Experimental): Standard therapy with Surgery, Temozolomide, and Radiotherapy; plus Trivax, 5x10e6 autologous interleukine-12 secreting dendritic cells charged with autologous tumour lysate.
  Interventions: Drug: Trivax, Temozolomide, Surgery, Radiotherapy
- Standard therapy (Active Comparator): Surgery, Temozolomide, Radiotherapy
  Interventions: Drug: Temozolomide, Surgery, Radiotherapy

INTERVENTIONS:
Drug: Trivax, Temozolomide, Surgery, Radiotherapy — Trivax: 5 x 10e6 dendritic cells, intranodal in 500 µl NaCl, weeks 7, 8, 9, 10, 12, 16, 20, 24, 28, 32
  Irradiation: 2 Gy per fraction once daily, five days per week (Mo-Fr), weeks 1, 2, 3, 4, 5, 6, total dose 60 Gy
  Temozolomide concomitant to radiotherapy: 75 mg/m²/day, 5 days per week (Mo-Fr), weeks 1, 2, 3, 4, 5, 6.
  Break: weeks 7, 8, 9, 10.
  Temozolomide adjuvant: 150 mg/m²/day, five days per week (Mo-Fr), week 11; 200 mg/m²/day, five days per week (Mo-Fr), weeks 15, 19, 23, 27, 31.
  Arms: Standard therapy plus Trivax
Drug: Temozolomide, Surgery, Radiotherapy — Irradiation: 2 Gy per fraction once daily, five days per week (Mo-Fr), weeks 1, 2, 3, 4, 5, 6, total dose 60 Gy
  Temozolomide concomitant to radiotherapy: 75 mg/m²/day, 5 days per week (Mo-Fr), weeks 1, 2, 3, 4, 5, 6
  Break: weeks 7, 8, 9, 10
  Temozolomide adjuvant: 150 mg/m²/day, five days per week (Mo-Fr), week 11; 200 mg/m²/day, five days per week (Mo-Fr), weeks 15, 19, 23, 27, 31
  Arms: Standard therapy

SUMMARY:
A randomised, open-label, 2-arm, multi-centre, phase II clinical study with one group receiving standard therapy with Temozolomide, radiotherapy, and Trivax; and a control group receiving standard therapy with Temozolomide and radiotherapy only; after tumour resection of at least 70% in both groups. The hypothesis is based on the assumption that time to progression will be doubled in the treatment group.

DETAILED DESCRIPTION:
Vaccination represents a success story in modern medicine and its principles have been found to be valid in different species, at least in the case of infectious diseases. As of today, there is little reason to believe that this would not be true in the case of tumours. It is now generally acknowledged that human tumours carry a mutational antigenic (non-self) repertoire of immunogenic potential that may be a suitable target for antitumour immune therapy. During the last years accumulating evidence from mouse experiments indicates that one can immunise prophylactically against cancers as effectively as against an infectious agent. However, in contrast to most experimental mouse tumour models, human tumours have in general been within their host for a long time and thus had the opportunity to influence their microenvironment and the larger immunological environment. Antigens capable of mediating specific rejection were found in human as well as in mouse tumours.

Many of the clinical trials using dendritic cell (DC) -based cancer vaccination techniques were designed for the treatment of melanoma. Other important diseases in which DC-based cancer vaccination was studied include prostate cancer, B cell lymphoma, renal cell carcinoma, glioma and glioblastoma, breast and ovarian cancer, gastrointestinal cancer, and selected solid paediatric tumours. In most of these trials some in vivo and/or in vitro evidence for the generation of anti-tumour immunity was found and even complete or partial remission of the tumour was observed in selected cases. The first phase III trial demonstrating the efficacy of DC cancer vaccination for the treatment of prostate cancer was reported recently (www.dendreon.com). Also patients suffering from glioblastoma multiforme appear to benefit from DC cancer immune therapy. The side effects observed in DC cancer vaccinations were usually described to be mild and not limiting the application.

We developed a DC cancer vaccine technology, Trivax, advancing the design of DC cancer immune therapy in one critical aspect. It is the first such vaccine that is enable for releasing the immune modulatory cytokine interleukin (IL) -12. Trivax is comprised of IL-12 secreting DCs and a mixture of protein tumour antigens derived from the individual patient's tumour cells. No synthetic tumour antigen component is involved. Both components of Trivax are derived from the individual patient and are used for the treatment of only this patient. Trivax therefore represents a fully individualised somatic cell therapy medicine. Trimed's early clinical evaluations in patients suffering from kidney cancer, prostate cancer, bone tumours, and malignancies of childhood have confirmed the safety and the feasibility of the Trivax technology.

Glioblastoma multiforme (GBM) (ICD-O M9440/3) is the most malignant astrocytic tumour, composed of poorly differentiated neoplastic astrocytes. Histopathological features include cellular polymorphism, nuclear atypia, brisk mitotic activity, vascular thrombosis, micro-vascular proliferation and necrosis. GBM typically affects patients of various age beginning in childhood and up to high age. It is preferentially located in the cerebral hemispheres. GBM may develop from diffuse astrocytomas WHO grade II or anaplastic astrocytomas (secondary GBM), but more frequently, they manifest after a short clinical history de novo, without evidence of a less malignant precursor lesion (primary GBM). In spite of modern oncological treatment, the prognosis of GBM remains dismal, with a median survival of little over 1 year.

GBM-Vax is a randomised, open-label, 2-arm, multi-centre, phase II clinical study with both groups undergoing surgery and receiving standard therapy with Temozolomide and radiotherapy; and the treatment group that in addition to the standard therapy receives cancer immune therapy with Trivax. Our aim is to extend therapy options presently including surgery, irradiation and Temozolomide with DC cancer vaccination to improve the poor prognosis of patients with GBM.

Primary objective

• Progression free survival measured as percentage of non-progressive patients with newly diagnosed GBM 12 months after a post-operative MRI scan treated according to the current standard (surgical resection, irradiation, oral chemo-therapy with Temozolomide), and Trivax, an autologous DC cancer vaccine charged with autologous tumour protein, as add-on therapy (group A), in comparison to patients receiving standard treatment without Trivax (group B).

Secondary objectives

* Progression free survival measured as percentage of non-progressive patients with newly diagnosed GBM 18 and 24 months after a post-operative MRI scan receiving standard treatment and Trivax as add-on therapy (group A), in comparison to patients receiving standard treatment without Trivax (group B).
* Extension of overall survival of patients with newly diagnosed GBM receiving standard treatment and Trivax as add-on therapy, in comparison to patients receiving standard treatment without Trivax.
* Quality of life in patients treated with Trivax as an add-on therapy using ECOG (Eastern Cooperative Oncology Group) performance status compared to qual-ity of life of patients receiving standard therapy (for study patients older 18 years).

Number of subjects In total, 56 patients will be enrolled in the study. The study consists of 2 arms and at least 28 patients should be randomly assigned to one of the two arms. It is expected to recruit the study patients within a period of one year. Randomisation is based on stratification according to study sites at a 1:1 ratio. Patients younger than 18 years will not be randomised but will all receive add-on therapy with Trivax. We feel that it would be not just to expect from children to understand and accept that there is a new treatment available but only every second patient will receive it. Obviously, patients younger than 18 years will not be analysed together with adult patients in the context of the study; and paediatric patients will not count towards the recruiting number of 2 x 28. Thus, the results obtained in paediatric GBM patients will not influence the outcome of the study in patients older than 18 years.

ELIGIBILITY:
Inclusion Criteria:

* Female or male, paediatric or adult patients of 3 to 70 years of age at time of diagnosis that qualify for standard treatment including surgery, Temozolomide and radiotherapy.
* GBM (WHO IV), confirmed by histology.
* Total, subtotal, or partial resection of more then 70% of tumour mass defined by MRI.
* Supratentorial tumour localisation.
* ECOG performance status 0, 1, or 2 (for study patients older 18 years).
* Life expectancy of at least 12 weeks by assessment of the attending physician.
* Written informed consent of patient and/or legal guardian in case of children or adolescents.

Exclusion Criteria:

* Less than 100 µg of tumour protein obtained from the resected tissue.
* Anti-neoplastic chemotherapy or radiotherapy during 4 weeks before entering the study, e.g. in another therapeutic phase I, II, or III study.
* Positive pregnancy test or breast-feeding.
* Patients unwilling to perform a save method of birth control.
* Known hypersensitivity to temozolomide.
* HIV positivity.

Ages: 3 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 87 (Actual)
Dates: Start 2010-04; Primary Completion 2015-06 (Actual); Study Completion 2015-11 (Actual)

PRIMARY OUTCOMES:
Progression free survival | 12 months
  Progression free survival measured as percentage of non-progressive patients with newly diagnosed GBM 12 months after a post-operative MRI scan treated according to the current standard (surgical resection, irradiation, oral chemotherapy with Temozolomide), and Trivax, an autologous DC cancer vaccine charged with autologous tumour protein, as add-on therapy (group A), in comparison to patients receiving standard treatment without Trivax (group B).

SECONDARY OUTCOMES:
Quality of Life | 24 months
  Quality of life in patients treated with Trivax as an add-on therapy using ECOG (Eastern Cooperative Oncology Group) performance status compared to quality of life of patients receiving standard therapy.
Progression free survival at 18 and 24 months | 24 months
  Progression free survival measured as percentage of non-progressive patients at 18 and 24 months post initiation of treat-ment.
Overall survival | 24 months
  The percentage of survival will be assessed at 12, 18, and 24 months.

CONTACTS AND LOCATIONS:
Overall Officials: Johanna Buchroithner, MD, Principal Investigator — Landesnervenklinik Wagner-Jauregg
Locations (8):
- Austria (8):
  - Landesnervenklinik Wagner-Jauregg, Linz, Upper Austria
  - Landeskrankenhaus Feldkirch, Feldkirch
  - Department of Neurosurgery, Medical University Graz, Graz
  - Clinical Department of Neurology, Medical University Innsbruck, Innsbruck
  - Department of Neurosurgery, Christian Doppler Klinik, Paracelsus Medizinische Privatuniversität, Salzburg
  - Neuroonkologisches Tumorboard KFJ-KA; Rudolfsstiftung, Vienna
  - Department of Paediatrics, Medical University Vienna, Vienna
  - Medical Department of Oncology, Donauspital, SMZ-Ost, Vienna

REFERENCES:
- [Background] Dohnal AM, Graffi S, Witt V, Eichstill C, Wagner D, Ul-Haq S, Wimmer D, Felzmann T. Comparative evaluation of techniques for the manufacturing of dendritic cell-based cancer vaccines. J Cell Mol Med. 2009 Jan;13(1):125-35. doi: 10.1111/j.1582-4934.2008.00304.x. Epub 2008 Mar 17. PMID 18363835
- [Background] Dohnal AM, Witt V, Hugel H, Holter W, Gadner H, Felzmann T. Phase I study of tumor Ag-loaded IL-12 secreting semi-mature DC for the treatment of pediatric cancer. Cytotherapy. 2007;9(8):755-70. doi: 10.1080/14653240701589221. Epub 2007 Oct 4. PMID 17917887
- [Background] Felzmann T, Huttner KG, Breuer SK, Wimmer D, Ressmann G, Wagner D, Paul P, Lehner M, Heitger A, Holter W. Semi-mature IL-12 secreting dendritic cells present exogenous antigen to trigger cytolytic immune responses. Cancer Immunol Immunother. 2005 Aug;54(8):769-80. doi: 10.1007/s00262-004-0637-2. Epub 2005 Jan 13. PMID 15647926
- [Background] Huttner KG, Breuer SK, Paul P, Majdic O, Heitger A, Felzmann T. Generation of potent anti-tumor immunity in mice by interleukin-12-secreting dendritic cells. Cancer Immunol Immunother. 2005 Jan;54(1):67-77. doi: 10.1007/s00262-004-0571-3. PMID 15693141
- [Background] Michael Dohnal A, Luger R, Paul P, Fuchs D, Felzmann T. CD40 ligation restores type 1 polarizing capacity in TLR4-activated dendritic cells that have ceased interleukin-12 expression. J Cell Mol Med. 2009 Aug;13(8B):1741-1750. doi: 10.1111/j.1582-4934.2008.00584.x. PMID 20187300
- [Background] Traxlmayr MW, Wesch D, Dohnal AM, Funovics P, Fischer MB, Kabelitz D, Felzmann T. Immune suppression by gammadelta T-cells as a potential regulatory mechanism after cancer vaccination with IL-12 secreting dendritic cells. J Immunother. 2010 Jan;33(1):40-52. doi: 10.1097/CJI.0b013e3181b51447. PMID 19952957